CLINICAL TRIAL: NCT06038240
Title: Optimizing Pain Self-Management in Total Knee Arthroplasty
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Patrick Finan, PhD, Harold Carron Professor, University of Virginia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HSR230005
Record Dates: First submitted 2023-09-07; First posted 2023-09-14 (Actual); Last update posted 2023-12-06 (Actual); Status verified 2023-11

CONDITIONS: Osteo Arthritis Knee; Knee Pain Chronic; Surgery
MeSH Terms: interventions — Educational Status

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Savoring Meditation (Experimental): A 4-session meditation intervention in which participants are trained to generate positive emotional states and focus their awareness on those states throughout the meditation.
  Interventions: Behavioral: Savoring Meditation
- Pain Self-Management and Education (Other): Education Control
  Interventions: Behavioral: Pain Self-Management and Education

INTERVENTIONS:
Behavioral: Savoring Meditation — Participants will learn about pain neuroscience and will learn/practice a positive emotion generative practice (Savoring Meditation).
  Arms: Savoring Meditation
Behavioral: Pain Self-Management and Education — Participants will learn about the biopsychosocial drivers of chronic pain.
  Arms: Pain Self-Management and Education

SUMMARY:
The purpose of this study is to investigate the efficacy of a positive affect enhancing intervention designed to reduce pain and augment reward system function in knee osteoarthritis (KOA) patients undergoing total knee arthroplasty (TKA). The scientific premise is that patient use of a positive emotion generative practice - savoring meditation, which has been demonstrated to reduce pain in experimental laboratory settings, enhanced with a pain neuroscience education component about reward system dysfunction as a chronic pain mechanism - is optimally suited to reduce postsurgical pain and augment reward system functioning relative to a Pain Self-Management and Education (PSME) condition. We will randomize 150 patients with KOA undergoing unilateral TKA to a brief, 4-session (20-30 minutes each) course of Savoring Meditation (SM; n = 75) or PSME (n = 75) delivered remotely by trained interventionists in a one-on-one format. We will assess pain and as well as pain-related risk and protective factors both via questionnaire and via weeklong ecological momentary assessment (EMA) data bursts on the following schedule: baseline, post-surgery, and 3-month follow-up. In addition, participants will attend laboratory testing sessions at baseline and 6-weeks post-surgery, during which affective pain modulation and electroencephalographic (EEG) brain biomarkers associated with pain and affect will be recorded. Participants in SM be encouraged to practice their savoring for 5 minutes/day during the week following surgery, as well as to use it to manage pain flares in a self-directed manner.

DETAILED DESCRIPTION:
Total knee arthroplasty (TKA) is an increasingly utilized, end-stage, cost-effective treatment for knee osteoarthritis (OA), one of the leading causes of disability worldwide whose hallmark symptoms include pain, stiffness, limited range of motion, and physical mobility limitations. The mechanisms of pain in OA, like most chronic pain conditions, are complex, multifaceted, and involve both central and peripheral sensitization , as well as reward system dysfunction. Despite its overall efficacy, a significant portion of patients with TKA (10-34%) continue to experience painful joints following the procedure , while an estimated 20% are dissatisfied with the outcome of their procedure. Further, an estimated 20% experience significant post-operative psychological distress in the months following surgery, which longitudinally predicts poorer functional outcomes. TKA on average fails to improve pain and function to a level comparable to the general population, or to the level achieved by other joint replacement procedures (i.e., hip arthroplasty) . These limitations highlight an urgent need to investigate safe and scalable strategies to improve TKA outcomes.

Psychosocial processes have a clinically meaningful role in shaping TKA outcomes. Well-established presurgical cognitive and affective risk factors include pain catastrophizing , kinesiophobia , poor outcome expectations and reward system dysfunction . Meanwhile, emerging research suggests that positive, resilience-related factors such as positive affect, vitality, vigor, social support, self-efficacy, and global, trait-like resilience predict more favorable TKA outcomes.

Major Gap in Knowledge

Despite known, modifiable psychological risk and resilience factors known to impact TKA outcomes, only recently have psychosocial processes in TKA been targeted in clinical trials. There are a handful of investigations which have variously employed psychoeducation, guided imagery, motivational interviewing, and cognitive-behavioral approaches, which have demonstrated modest to poor efficacy in impacting postsurgical pain and function. Pain neuroscience education (PNE) is a relatively recent psychosocial intervention approach to chronic pain that educates patients on the modern neuroscientific understanding of mechanisms (e.g., central and peripheral sensitization), whose efficacy appears to be optimized when combined with an additional active treatment (e.g., physical therapy) informed by the patent's reconceptualization of pain (away from biomedical or biomechanical understanding and towards a modern neuroscientific understanding) achieved through PNE. Initial studies on PNE alone in TKA patients show a favorable effect on patient satisfaction with the TKA procedure and psychosocial risk factors including pain catastrophizing and kinesiophobia but no effect on pain or function.

How Proposed Work Will Fill the Gaps

The present study will address major gaps in knowledge by testing a novel prophylactic psychological intervention for TKA patients that targets reward system dysfunction, a central driver of chronic pain states. Specifically, the study will test a novel Savoring Meditation (SM) intervention, which teaches patients how to augment positive affective functioning via meditating on a positive autobiographical memory. In addition, using a pain neuroscience education framework, SM will also educate participants on the neurophysiological basis for engaging in savoring meditation. Specifically, the intervention will educate patients about the reward system in the brain, and how deficits in reward system functioning serve to maintain pain. Subsequently, the intervention will explain to patients that savoring meditation has been empirically shown and is optimally suited to reduce pain vis-a-vis augmented reward system functioning. Patients randomized to SM will engage in 4 sessions of SM with a trained interventionist. They will be encouraged to use their SM skills in the postsurgical period to manage pain. The study will compare the efficacy of SM to a Pain Self-Management and Education (PSME) condition, wherein patients will learn about biological, psychological, and social drivers of pain. The PSME condition will control for therapeutic alliance and treatment expectancies. It is hypothesized that patients who undergo 4 sessions of SM will demonstrate reduced clinical pain and prescription opioid use across major assessment timepoints (post-treatment, 6-weeks, and 3-months), relative to PSME. Reward system function measured via self-report, affective pain modulation task performance, and electroencephalographic (EEG) based biomarkers will be investigated as a secondary outcome.

ELIGIBILITY:
Inclusion Criteria:

* 18-85 years old.
* Have a physician-confirmed treatment plan to undergo unilateral TKA along with physician-confirmed knee osteoarthritis diagnosis.
* Willingness and ability to comply with scheduled sessions and study procedures

Exclusion Criteria:

* Member of a vulnerable population including pregnant women, children, prisoners, cognitively impaired, and non-English-speaking subjects.
* Current unstable, severe medical comorbidity.
* Current severe psychiatric comorbidity (e.g., schizophrenia, psychosis, or other unstable psychiatric disorder).
* Current severe alcohol or substance use disorder.
* Weekly or more frequent use of opioids in the past 30 days (other than tramadol and/or codeine) for therapeutic or non-therapeutic purposes.
* Other surgery of the affected knee in the last 6 months.
* Previous TKA.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2023-11-27 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Numeric Rating Scale for Clinical Pain | Baseline to 3 months post-surgery
  Average pain intensity on numeric rating scale (range of 0-100; higher scores indicate greater pain), aggregated across Ecological Momentary Assessment observations
Opioid Use | Baseline to 3-months post-surgery
  Morphine Equivalent Units per day, as assessed with Ecological Momentary Assessment

SECONDARY OUTCOMES:
Knee Injury and Osteoarthritis Outcome Score for Joint Replacement (KOOS JR) | Baseline to 3 months post-surgery
  Measure of pain and function following knee surgery (range of 1-100; higher scores indicate higher level of function)
Positive and Negative Outcome Schedule-X (PANAS-X) Joviality Subscale | Baseline to 3-months post-surgery
  Measure of positive emotion (range of 1-5; higher scores indicate greater positive emotion)
Snaith-Hamilton Pleasure Scale (SHAPS) | Baseline to 3-months post-surgery
  Measure of anhedonia (range of 14-56; higher scores indicate greater anhedonia)

CONTACTS AND LOCATIONS:
Locations (1):
- Fontaine Research Park, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified data will be shared upon reasonable request from other researchers, and after a data use agreement has been executed between institutions.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Data will become available after the study is complete and the primary outcomes manuscript has been published.
Access Criteria: Access will be granted after a Data Use Agreement has been executed.